CLINICAL TRIAL: NCT03979404
Title: A Feasibility Case Series of Theta Burst Stimulation in Anorexia Nervosa
Brief Title: Theta Burst Stimulation in Anorexia Nervosa: A Case Series
Acronym: ANTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCLANTSCASE19
Record Dates: First submitted 2019-06-04; First posted 2019-06-07 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Anorexia Nervosa
Keywords: Theta Burst Stimulation; Neuromodulation; Psychiatric Disorders; Transcranial Magnetic Stimulation; Anorexia Nervosa; Eating Disorders
MeSH Terms: conditions — Anorexia Nervosa; Mental Disorders; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active iTBS (Experimental): iTBS will be delivered at 80% of resting motor threshold, consisting of a triplet of 50Hz bursts, repeated at 5Hz; 2 seconds on and 8 seconds off; 600 pulses per session; total duration of 3 minutes and 9 seconds, to the left dorsolateral prefrontal cortex.
  Interventions: Device: Intermittent Theta Burst Stimulation

INTERVENTIONS:
Device: Intermittent Theta Burst Stimulation — The Magstim Rapid2 Magnetic Stimulator (Magstim ®, UK) will be used to administer active TBS.
  Other Names: iTBS

SUMMARY:
Anorexia Nervosa (AN) is a life-threatening eating disorder characterised by an intense fear of weight gain and disturbed body image, which motivates severe dietary restriction or other weight loss behaviours (e.g. purging). Treatment efficacy in adults with AN remains low: only a small percentage of individuals fully recover, and dropout rates are high. For adolescents with a relatively short term illness duration (under 3 years), family-based therapy has been associated with more favourable outcomes. However, for those adolescents with a longer illness duration (over 3 years), there are no specific treatments associated with positive long-term outcomes and these individuals are at risk of developing a severe and enduring form of the illness (SE-AN).

In part, treatment can be problematic due to ambivalence, which is reflected in poor take-up of certain treatments (e.g. pharmacological treatments that lead to weight gain) and high drop-out rates. Repetitive transcranial magnetic stimulation (rTMS) has demonstrated efficacy for treatment of AN in adults and improving treatment adherence. However, this has yet to be investigated in adolescents with AN.

This study will use a novel type of rTMS, called intermittent theta burst stimulation (iTBS). TBS takes as little as a few minutes duration compared to the classical rTMS protocol which takes approximately 37.5 minutes. In addition, TBS has been found to produce longer after-effects of the induced plastic changes and has a lower stimulation intensity, which may therefore be more practical and potentially safer to administer in people with AN. Thus, the aim of this feasibility case series is to obtain preliminary data on the longer-term (i.e. up to 6 months) effects of 20 sessions of iTBS on reducing core symptoms of AN.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants over the age of 13
* BMI over 14 (for participants over the age of 18) or over 66% of the median BMI for age and gender (for participants under the age of 18)
* Right-handed
* Current Diagnostic and Statistical Manual-5 (DSM-5) diagnosis of AN-restricting type (AN-R) or AN-binge/purge type (AN-BP) and an illness duration of 3 years or more
* Must have completed at least one adequate previous course of eating disorder treatment (e.g. one 6-month course of specialist outpatient therapy, specialist day-care or in-patient treatment for refeeding)
* Participants under the age of 18 must have informed consent from parent(s)/carer(s)
* Must have approval from treating eating disorders clinician or general practitioner (GP) to participate

Exclusion Criteria:

* Having a history of head or eye injury
* Having a history of a neurological disease including previous seizures of any kind
* Having metallic implants anywhere in the head or body
* Being on a dose of any psychotropic medication that has not been stable for at least 14 days prior to participation in the study
* Taking antipsychotic medication
* Taking anti-convulsive medication
* Pregnancy or suspected pregnancy in female participants
* Having a current other major psychiatric disorder (e.g. major depressive disorder, substance dependence, schizophrenia or bipolar) needing treatment in its own right
* Excessive alcohol (>3 units per day, 5 days of the week) and/or cigarette consumption (>15 cigarettes per day)
* Severe abnormalities in the screening clinical blood sample
* An rTMS safety questionnaire and an MRI safety questionnaire will also be administered and if deemed not safe to deliver rTMS or undergo MRI scanning, people will be excluded on this basis.

Ages: 13 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-02-18 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Changes in core symptoms of AN from baseline to post-treatment | Throughout the study, lasting 7 months: baseline (before treatment), weekly throughout 4-weeks of treatment and 6 months after treatment (long-term follow-up)
  Core symptoms of AN are computed by summing scores on three 10cm visual analogue scales (maximum score of 30) that assess levels of "urge to restrict", "feeling full", and "feeling fat". Participants are requested to indicate on this line a degree or level of experiencing the specific emotion or behavioural urge from "not at all" to "severe".

SECONDARY OUTCOMES:
Changes in performance on the Two-step Sequential Learning Task from baseline to post-treatment | 1 month: baseline (before treatment) and post-treatment
  Neuropsychological task measuring model-based and model-free reinforcement learning
Changes in performance on the Food Choice Task from baseline to post-treatment | 1 month: baseline (before treatment) and post-treatment
  Neuropsychological task measuring decision making regarding food selection
Changes in performance on the Face Affective Go No-Go Task from baseline to post-treatment | 1 month: baseline (before treatment) and post-treatment
  Neuropsychological task measuring information processing biases for positive and negative facial expressions
Changes in performance on the Visual Probe Task from baseline to post-treatment | 1 month: baseline (before treatment) and post-treatment
  Neuropsychological task measuring information processing biases to high and low calorie foods
Changes in performance on the Emotion Regulation Task from baseline to post-treatment | 1 month: baseline (before treatment and post-treatment
  Neuropsychological task measuring heart rate variability (as an index of autonomic nervous system activity) during presentation of highly aversive pictures
Changes in self-reported perception of low mood from baseline to post-treatment | 7 months: baseline (before treatment), post-treatment and at 6-month follow-up (long-term follow-up)
  Low mood is measured on a 10cm visual analogue scale (maximum score 10). Participants are requested to indicate on this line a degree or level of experiencing "low mood" from "not at all" to "severe". Therefore a higher score reflects higher feelings of low mood.
Changes in self-reported perception of anxiety from baseline to post-treatment | 7 months: baseline (before treatment), post-treatment and at 6-month follow-up (long-term follow-up)
  Anxiety is measured on a 10cm visual analogue scale (maximum score 10). Participants are requested to indicate on this line a degree or level of experiencing "anxiety" from "not at all" to "severe". Therefore a higher score reflects higher feelings of anxiety.
Changes in self-reported perception of urge to exercise from baseline to post-treatment | 7 months: baseline (before treatment), post-treatment and at 6-month follow-up (long-term follow-up)
  Urge to exercise is measured on a 10cm visual analogue scale (maximum score 10). Participants are requested to indicate on this line a degree or level of experiencing "urge to exercise" from "not at all" to "severe". Therefore a higher score reflects a higher urge to exercise.
Changes in self-reported perception of urge to be sick/purge from baseline to post-treatment | 7 months: baseline (before treatment), post-treatment and at 6-month follow-up (long-term follow-up)
  Urge to be sick/purge is measured on a 10cm visual analogue scale (maximum score 10). Participants are requested to indicate on this line a degree or level of experiencing "urge to be sick/purge" from "not at all" to "severe". Therefore a higher score reflects a higher urge to be sick/purge.
Changes in global scores on the Depression and Anxiety Stress Scale (DASS-21) from baseline to post-treatment | 7 months: baseline (before treatment), post-treatment and at 6-month follow-up (long-term follow-up)
  The DASS-21 is a self-report questionnaire of 21 items, 7 items per sub-scale: depression, anxiety and stress. Participants are asked to score every item on a scale from 0 (did not apply to me at all) to 3 (applied to me very much) based on how much each statement applies to them over the past week. Global score is computed by adding up the scores on the items per sub-scale and multiplying them by a factor 2, therefore higher scores reflecting more severe depressive symptoms. Global scores for the DASS-21 range between 0 and 120.
Changes in global scores on the Eating Disorder Examination Questionnaire (EDE-Q) from baseline to post-treatment | 7 months: baseline (before treatment), post-treatment and at 6-month follow-up (long-term follow-up)
  The EDE-Q is a 28-item questionnaire that provides a measure of the range and severity of eating disorder features experienced over the past 28 days. The EDE-Q is scored using a 7-point, forced-choice rating scale (0-6) with higher scores reflecting a higher level of symptomatology. The EDE-Q yields a global score and four sub-scale scores: restraint, shape concern, weight concern, eating concern. The global score is calculated as the sum of the four sub-scale scores divided by the number of sub-scales (i.e. four). Global scores for the EDE-Q range between 0 and 6.
Changes in body mass index (BMI; kg/m2) from baseline to post-treatment | 7 months: baseline (before treatment), post-treatment and at 6-month follow-up (long-term follow-up)
  BMI is a simple calculation of a person's height (m2; metres squared) and weight (kilograms). It is widely used as a general indicator of whether a person has a healthy body weight for their height.

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom